CLINICAL TRIAL: NCT01592240
Title: A Phase 2b Double-blind, Randomized, Placebo-controlled, Parallel Group, Dose-ranging Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 Following Monthly And Twice Monthly Subcutaneous Dosing For Six Months In Hypercholesterolemic Subjects On A Statin
Brief Title: Monthly And Twice Monthly Subcutaneous Dosing Of PF-04950615 (RN316) In Hypercholesterolemic Subjects On A Statin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1481015; 2012-001226-10 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Hypercholesterolemia
Keywords: PF-04950615; RN316
MeSH Terms: conditions — Hypercholesterolemia | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q28d Dosing Arm (Experimental): A total of 7 dose groups in two dosing schedules, 50 subjects per dose group are planned. Q28d dose group will receive subcutaneous administration of PF-04950615 or Placebo once a month.
  Interventions: Drug: PBO; Drug: 200mg PF-04950615 (RN316); Drug: 300mg PF-04950615 (RN316)
- Q14d Dosing Arm (Experimental): A total of 7 dose groups in two dosing schedules, 50 subjects per dose group are planned. Q14d dose group will receive subcutaneous administration of PF-04950615 or Placebo every 2 weeks.
  Interventions: Drug: PBO; Drug: PF-04950615

INTERVENTIONS:
Drug: PBO — Placebo Q28d
  Arms: Q28d Dosing Arm
Drug: 200mg PF-04950615 (RN316) — PF-04950615 200 mg, Q28d
  Other Names: PF-04950615 (RN316)
  Arms: Q28d Dosing Arm
Drug: 300mg PF-04950615 (RN316) — PF-04950615 300 mg, Q28d
  Other Names: PF-04950615 (RN316)
  Arms: Q28d Dosing Arm
Drug: PBO — Placebo, Q14d
  Arms: Q14d Dosing Arm
Drug: PF-04950615 — PF-04950615 50mg, Q14d
  Other Names: PF-04950615 (RN316)
  Arms: Q14d Dosing Arm
Drug: PF-04950615 — PF-04950615 100 mg, Q14d
  Other Names: PF-04950615 (RN316)
  Arms: Q14d Dosing Arm
Drug: PF-04950615 — PF-04950615 150mg, Q14d
  Other Names: PF-04950615 (RN316)
  Arms: Q14d Dosing Arm

SUMMARY:
To evaluate the Low Density Lipoprotein-Cholesterol (LDL-C) lowering effect of PF-04950615 administered subcutaneously at monthly intervals, or twice monthly intervals in subjects with high cholesterol whose LDL-cholesterol is >/=80 mg/dL on background treatment with a statin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be receiving a stable dose (at least 6 weeks) of any statin and continue on same dose of statin for the duration of this trial.
* Lipids should meet the following criteria on a background treatment with a statin at 2 screening visits that occur at screening and at least 7 days prior to randomization on Day 1:
* Fasting LDL-C greater than or equal to 80 mg/dL (2.31 mmol/L);
* Fasting TG less than or equal to 400 mg/dL (4.52 mmol/L).
* Subject's fasting LDL-cholesterol must greater than or equal to 80 mg/dL (2.31 mmol/L at the initial screening visit, and the value at the second visit within 7 days of randomization must be not lower than 20% of this initial value to meet eligibility criterion for this trial.

Exclusion Criteria:

* Participation in other studies within 3 months before the current study begins and/or during study participation.
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Pregnant females; breastfeeding females; males and females of childbearing potential not using highly effective contraception or not agreeing to continue highly effective contraception for at least 63 days after last dose of investigational product.
* History of a cardiovascular or cerebrovascular event or procedure (eg, MI, stroke, TIA, angioplasty) during the past 6 months. Congestive heart failure (CHF), NYHA functional classes III or IV.
* Poorly controlled type 1 or type 2 diabetes mellitus (defined as HbA1c >9%).
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- United States (74):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - The Office of James G. McMurray, MD, Huntsville, Alabama
  - Southwest Heart Group, Tucson, Arizona
  - Aureus Research Inc., Little Rock, Arkansas
  - Universal Biopharma Research Institute Inc. - Alta Family Health Clinic, Dinuba, California
  - Clinical Trials Research, Lincoln, California
  - The Office of Lucita M. Cruz, MD, Inc., Norwalk, California
  - Radiant Research, Santa Rosa, California
  - St. Joseph's Medical Associates, Stockton, California
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Zasa Clinical Research, Boynton Beach, Florida
  - Florida Health Center, Davie, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - In Vivo Clinical Research, Inc., Hialeah, Florida
  - Health Care Family Rehab and Research Center, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Community Research Foundation, Inc., Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - DMI Research, Pinellas Park, Florida
  - St Johns Center for Clinical Research, Ponte Vedra, Florida
  - The Office of Bridget Bellingar, DO, Seminole, Florida
  - Miami Research Associates, South Miami, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Radiant Research, Inc., Atlanta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Northwest Clinical Trials, Boise, Idaho
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Radiant Research, Inc., Chicago, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Midwest Heart & Vascular Specialists, Overland Park, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Maine Research Associates, Lewiston, Maine
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Radiant Research, Inc., Edina, Minnesota
  - Dybedal Clinical Research Center, Kansas City, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Meridian Clinical Research, Omaha, Nebraska
  - New Mexico Clinical Research and Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Central New York Clinical Research, Manlius, New York
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - Wake Internal Medicine Consultants, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - Clinical Trials of America, Inc., Winston-Salem, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Sterling Research Group, LTD., Cincinnati, Ohio
  - Albert J. Weisbrot, M.D., Inc., Mason, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Baylor College of Medicine - Center for Cardiovascular Disease Prevention, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - National Clinical Research- Norfolk, Inc, Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Ballantyne CM, Neutel J, Cropp A, Duggan W, Wang EQ, Plowchalk D, Sweeney K, Kaila N, Vincent J, Bays H. Results of bococizumab, a monoclonal antibody against proprotein convertase subtilisin/kexin type 9, from a randomized, placebo-controlled, dose-ranging study in statin-treated subjects with hypercholesterolemia. Am J Cardiol. 2015 May 1;115(9):1212-21. doi: 10.1016/j.amjcard.2015.02.006. Epub 2015 Feb 12. PMID 25784512
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481015&StudyName=Monthly%20And%20Twice%20Monthly%20Subcutaneous%20Dosing%20Of%20PF-04950615%20%28RN316%29%20%20In%20Hypercholesterolemic%20Subjects%20On%20A%20Statin

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Every 14 Days: Participants received single dose of subcutaneous (SC) injection of placebo matched to PF-04950615 once every 14 days for 24 weeks.
- PF-04950615 50 mg: Every 14 Days: Participants received single dose of SC injection of PF-04950615 50 milligram (mg) once every 14 days for 24 weeks.
- PF-04950615 100 mg: Every 14 Days: Participants received single dose of SC injection of PF-04950615 100 mg once every 14 days for 24 weeks.
- PF-04950615 150 mg: Every 14 Days: Participants received single dose of SC injection of PF-04950615 150 mg once every 14 days for 24 weeks.
- Placebo: Every 28 Days: Participants received single dose of SC injection of placebo matched to PF-04950615 once every 28 days for 24 weeks.
- PF-04950615 200 mg: Every 28 Days: Participants received single dose of SC injection of PF-04950615 200 mg once every 28 days for 24 weeks.
- PF-04950615 300 mg: Every 28 Days: Participants received single dose of SC injection of PF-04950615 300 mg once every 28 days for 24 weeks.
Period: Overall Study
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Started | 50 | 50 | 52 | 50 | 51 | 50 | 51
Completed | 47 | 39 | 45 | 47 | 44 | 47 | 48
Not Completed | 3 | 11 | 7 | 3 | 7 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1 | 0 | 3 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 4 | 1 | 3 | 0 | 2
Not completed — Other | 0 | 3 | 1 | 1 | 0 | 0 | 1
Not completed — Did Not Meet Entrance Criteria | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days | Total
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51 | 354
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.84) | 59.1 (11.26) | 61.9 (9.58) | 61.4 (9.75) | 58.4 (11.62) | 60.3 (9.64) | 60.2 (8.17) | 60.3 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 26 | 29 | 22 | 31 | 26 | 185
  Male | 25 | 24 | 26 | 21 | 29 | 19 | 25 | 169

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: Full analysis set included all participants who were randomized. Here "Overall Number of Participants Analyzed", signifies number of participants those who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 47 | 44 | 42 | 46 | 46 | 48 | 50
milligram per deciliter (mg/dL) | -2.6 [-10.14 to 4.98] | -36.9 [-44.55 to -29.17] | -47.6 [-55.45 to -39.85] | -56.0 [-63.60 to -48.40] | 4.6 [-4.59 to 13.73] | -23.0 [-32.00 to -14.02] | -40.3 [-49.09 to -31.48]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -34.28, 95% CI 2-sided [-45.06 to -23.50]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -45.07, 95% CI 2-sided [-55.93 to -34.21]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -53.42, 95% CI 2-sided [-64.14 to -42.70]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -27.58, 95% CI 2-sided [-40.49 to -14.67]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -44.85, 95% CI 2-sided [-57.65 to -32.05]

2. Secondary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 48
milligram per deciliter | -3.6 [-11.16 to 3.88] | -32.0 [-39.72 to -24.37] | -46.8 [-54.44 to -39.25] | -44.7 [-52.19 to -37.16] | -0.6 [-7.69 to 6.54] | -24.3 [-31.21 to -17.49] | -30.9 [-37.71 to -24.18]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -28.41, 95% CI 2-sided [-39.15 to -17.67]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -43.21, 95% CI 2-sided [-53.90 to -32.51]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -41.03, 95% CI 2-sided [-51.66 to -30.41]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -23.77, 95% CI 2-sided [-33.70 to -13.84]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -30.36, 95% CI 2-sided [-40.24 to -20.49]

3. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: Full analysis set included all participants who were randomized. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 44 | 42 | 46 | 46 | 48 | 50
  Percent Change at Week 12 | 0.6 [-6.34 to 7.54] | -34.4 [-41.47 to -27.34] | -41.7 [-48.90 to -34.54] | -52.5 [-59.51 to -45.54] | 6.7 [-1.30 to 14.73] | -20.2 [-28.10 to -12.39] | -34.4 [-42.11 to -26.72]
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 48
  Percent Change at Week 24 | -0.9 [-7.39 to 5.64] | -30.0 [-36.64 to -23.29] | -41.0 [-47.62 to -34.42] | -40.0 [-46.55 to -33.51] | 2.4 [-4.08 to 8.96] | -21.3 [-27.63 to -15.07] | -26.6 [-32.84 to -20.45]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -35.00, 95% CI 2-sided [-44.91 to -25.10]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -42.32, 95% CI 2-sided [-52.30 to -32.33]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -53.12, 95% CI 2-sided [-62.97 to -43.27]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -26.96, 95% CI 2-sided [-38.25 to -15.67]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -41.13, 95% CI 2-sided [-52.32 to -29.94]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -29.09, 95% CI 2-sided [-38.42 to -19.77]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -40.14, 95% CI 2-sided [-49.43 to -30.86]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -39.16, 95% CI 2-sided [-48.37 to -29.94]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -23.79, 95% CI 2-sided [-32.88 to -14.70]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -29.08, 95% CI 2-sided [-38.13 to -20.04]

4. Secondary Outcome: Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 43 | 44 | 46 | 47 | 48 | 50
  Change at Week 12 | 0.3 [-1.80 to 2.39] | 1.9 [-0.20 to 4.06] | 2.0 [-0.08 to 4.13] | 0.8 [-1.28 to 2.92] | -1.0 [-3.33 to 1.27] | 3.4 [1.12 to 5.72] | 2.8 [0.58 to 5.08]
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Change at Week 24 | -0.2 [-2.09 to 1.79] | 1.6 [-0.44 to 3.57] | 0.6 [-1.32 to 2.61] | 0.3 [-1.60 to 2.28] | 0.2 [-2.39 to 2.72] | 2.2 [-0.32 to 4.66] | 0.2 [-2.28 to 2.60]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.281, Mixed models repeated measures analysis; Adjusted Mean Difference = 1.64, 95% CI 2-sided [-1.35 to 4.63]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.251, Mixed models repeated measures analysis; Adjusted mean difference = 1.73, 95% CI 2-sided [-1.24 to 4.71]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.724, Mixed models repeated measures analysis; Adjusted mean difference = 0.53, 95% CI 2-sided [-2.43 to 3.50]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.007, Mixed models repeated measures analysis; Adjusted mean difference = 4.45, 95% CI 2-sided [1.21 to 7.70]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.019, Mixed models repeated measures analysis; Adjusted mean difference = 3.86, 95% CI 2-sided [0.63 to 7.09]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.225, Mixed models repeated measures analysis; Adjusted mean difference = 1.72, 95% CI 2-sided [-1.07 to 4.51]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.571, Mixed models repeated measures analysis; Adjusted mean difference = 0.79, 95% CI 2-sided [-1.97 to 3.56]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.725, Mixed models repeated measures analysis; Adjusted mean difference = 0.49, 95% CI 2-sided [-2.25 to 3.24]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.268, Mixed models repeated measures analysis; Adjusted mean difference = 2.01, 95% CI 2-sided [-1.56 to 5.57]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.996, Mixed models repeated measures analysis; Adjusted mean difference = -0.01, 95% CI 2-sided [-3.55 to 3.54]

5. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 43 | 44 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | 1.2 [-2.87 to 5.25] | 4.6 [0.48 to 8.74] | 3.8 [-0.27 to 7.89] | 2.5 [-1.52 to 6.61] | -0.4 [-4.91 to 4.06] | 7.2 [2.76 to 11.72] | 6.1 [1.71 to 10.50]
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | -0.3 [-4.07 to 3.55] | 3.6 [-0.27 to 7.55] | 0.6 [-3.26 to 4.43] | 2.3 [-1.49 to 6.11] | 1.7 [-2.79 to 6.14] | 4.7 [0.34 to 8.99] | 1.0 [-3.27 to 5.22]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.246, Mixed models repeated measures analysis; Adjusted mean difference = 3.41, 95% CI 2-sided [-2.38 to 9.21]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.371, Mixed models repeated measures analysis; Adjusted mean difference = 2.62, 95% CI 2-sided [-3.14 to 8.38]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.643, Mixed models repeated measures analysis; Adjusted mean difference = 1.35, 95% CI 2-sided [-4.40 to 7.10]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.018, Mixed models repeated measures analysis; Adjusted mean difference = 7.66, 95% CI 2-sided [1.33 to 13.99]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.043, Mixed models repeated measures analysis; Adjusted mean difference = 6.52, 95% CI 2-sided [0.22 to 12.83]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.160, Mixed models repeated measures analysis; Adjusted mean difference = 3.90, 95% CI 2-sided [-1.56 to 9.36]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.758, Mixed models repeated measures analysis; Adjusted mean difference = 0.85, 95% CI 2-sided [-4.56 to 6.25]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.347, Mixed models repeated measures analysis; Adjusted mean difference = 2.57, 95% CI 2-sided [-2.81 to 7.95]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.343, Mixed models repeated measures analysis; Adjusted mean difference = 2.99, 95% CI 2-sided [-3.22 to 9.21]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.824, Mixed models repeated measures analysis; Adjusted mean difference = -0.70, 95% CI 2-sided [-6.87 to 5.48]

6. Secondary Outcome: Change From Baseline in Apolipoprotein B (ApoB) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Change at Week 12 | -2.8 [-7.65 to 2.02] | -21.4 [-26.26 to -16.48] | -30.5 [-35.40 to -25.57] | -34.9 [-39.77 to -30.04] | 2.3 [-3.59 to 8.24] | -12.2 [-18.08 to -6.40] | -26.2 [-31.92 to -20.42]
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 47 | 49 | 43
  Change at Week 24 | -2.5 [-7.68 to 2.66] | -22.2 [-27.46 to -16.89] | -30.7 [-35.92 to -25.44] | -27.9 [-33.09 to -22.75] | -2.9 [-7.70 to 1.83] | -15.7 [-20.26 to -11.06] | -19.8 [-24.32 to -15.26]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted Mean Difference = -18.55, 95% CI 2-sided [-25.44 to -11.67]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -27.67, 95% CI 2-sided [-34.55 to -20.79]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -32.09, 95% CI 2-sided [-38.95 to -25.22]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -14.56, 95% CI 2-sided [-22.89 to -6.24]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -28.50, 95% CI 2-sided [-36.83 to -20.16]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -19.67, 95% CI 2-sided [-27.07 to -12.27]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -28.17, 95% CI 2-sided [-35.52 to -20.82]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -25.41, 95% CI 2-sided [-32.73 to -18.09]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -12.72, 95% CI 2-sided [-19.35 to -6.09]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -16.85, 95% CI 2-sided [-23.47 to -10.23]

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | -1.9 [-7.31 to 3.45] | -23.5 [-28.94 to -18.07] | -32.5 [-37.93 to -27.01] | -37.9 [-43.29 to -32.47] | 3.7 [-2.55 to 9.86] | -13.5 [-19.60 to -7.37] | -27.1 [-33.09 to -21.04]
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | -1.5 [-7.27 to 4.25] | -23.6 [-29.48 to -17.72] | -32.5 [-38.29 to -26.64] | -28.7 [-34.50 to -22.99] | -1.4 [-6.88 to 3.98] | -16.8 [-22.04 to -11.54] | -20.6 [-25.76 to -15.42]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -21.58, 95% CI 2-sided [-29.23 to -13.92]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -30.54, 95% CI 2-sided [-38.19 to -22.89]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -35.95, 95% CI 2-sided [-43.59 to -28.31]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -17.14, 95% CI 2-sided [-25.87 to -8.41]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -30.72, 95% CI 2-sided [-39.45 to -21.98]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -22.09, 95% CI 2-sided [-30.32 to -13.86]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -30.95, 95% CI 2-sided [-39.13 to -22.77]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -27.23, 95% CI 2-sided [-35.38 to -19.09]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -15.34, 95% CI 2-sided [-22.90 to -7.78]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p < 0.001, Mixed models repeated measures analysis; Adjusted mean difference = -19.15, 95% CI 2-sided [-26.70 to -11.59]

8. Secondary Outcome: Change From Baseline in Apolipoprotein A1 (ApoA1) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Change at Week 12 | 2.1 [-3.56 to 7.85] | 3.9 [-1.83 to 9.67] | 7.6 [1.84 to 13.33] | 6.0 [0.25 to 11.68] | 2.2 [-2.37 to 6.84] | 7.8 [3.24 to 12.43] | 6.6 [2.09 to 11.11]
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Change at Week 24 | 0.8 [-4.59 to 6.12] | 1.4 [-4.14 to 6.86] | 1.2 [-4.19 to 6.58] | 4.9 [-0.45 to 10.23] | 2.0 [-3.76 to 7.72] | 0.6 [-5.01 to 6.15] | -0.2 [-5.68 to 5.26]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.667, Mixed models repeated measures analysis; Adjusted Mean Difference = 1.77, 95% CI 2-sided [-6.33 to 9.88]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.187, Mixed models repeated measures analysis; Adjusted mean difference = 5.44, 95% CI 2-sided [-2.66 to 13.54]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.352, Mixed models repeated measures analysis; Adjusted mean difference = 3.82, 95% CI 2-sided [-4.25 to 11.90]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.090, Mixed models repeated measures analysis; Adjusted mean difference = 5.60, 95% CI 2-sided [-0.89 to 12.09]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.184, Mixed models repeated measures analysis; Adjusted mean difference = 4.36, 95% CI 2-sided [-2.10 to 10.82]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.879, Mixed models repeated measures analysis; Adjusted mean difference = 0.59, 95% CI 2-sided [-7.09 to 8.28]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.911, Mixed models repeated measures analysis; Adjusted mean difference = 0.43, 95% CI 2-sided [-7.17 to 8.02]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.283, Mixed models repeated measures analysis; Adjusted mean difference = 4.12, 95% CI 2-sided [-3.44 to 11.69]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.728, Mixed models repeated measures analysis; Adjusted mean difference = -1.41, 95% CI 2-sided [-9.41 to 6.59]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.587, Mixed models repeated measures analysis; Adjusted mean difference = -2.19, 95% CI 2-sided [-10.13 to 5.75]

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A1 (ApoA1) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | 2.6 [-4.06 to 9.28] | 2.0 [-4.65 to 8.55] | 4.9 [-1.63 to 11.48] | 9.1 [2.52 to 15.77] | 2.2 [-0.84 to 5.24] | 5.7 [2.67 to 8.74] | 4.9 [1.90 to 7.85]
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | 1.4 [-3.65 to 6.44] | 0.5 [-4.53 to 5.59] | 0.2 [-4.73 to 5.22] | 7.2 [2.20 to 12.22] | 1.9 [-1.86 to 5.56] | 1.0 [-2.58 to 4.62] | 0.3 [-3.23 to 3.83]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.890, Mixed models repeated measures analysis; Adjusted mean difference = -0.66, 95% CI 2-sided [-10.05 to 8.74]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.625, Mixed models repeated measures analysis; Adjusted mean difference = 2.32, 95% CI 2-sided [-7.04 to 11.68]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.172, Mixed models repeated measures analysis; Adjusted mean difference = 6.54, 95% CI 2-sided [-2.86 to 15.94]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.109, Mixed models repeated measures analysis; Adjusted mean difference = 3.50, 95% CI 2-sided [-0.79 to 7.80]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.218, Mixed models repeated measures analysis; Adjusted mean difference = 2.67, 95% CI 2-sided [-1.60 to 6.94]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.812, Mixed models repeated measures analysis; Adjusted mean difference = -0.86, 95% CI 2-sided [-8.01 to 6.29]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.749, Mixed models repeated measures analysis; Adjusted mean difference = -1.15, 95% CI 2-sided [-8.24 to 5.94]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.108, Mixed models repeated measures analysis; Adjusted mean difference = 5.82, 95% CI 2-sided [-1.29 to 12.93]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.752, Mixed models repeated measures analysis; Adjusted mean difference = -0.83, 95% CI 2-sided [-5.99 to 4.34]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.550, Mixed models repeated measures analysis; Adjusted mean difference = -1.55, 95% CI 2-sided [-6.68 to 3.57]

10. Secondary Outcome: Change From Baseline in Apolipoprotein AII (ApoAII) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Change at Week 12 | 1.0 [-0.99 to 2.95] | 1.2 [-0.84 to 3.18] | 2.3 [0.29 to 4.32] | 0.3 [-1.65 to 2.33] | 1.7 [-0.20 to 3.65] | 1.2 [-0.67 to 3.13] | 2.1 [0.25 to 4.01]
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 46 | 43 | 47 | 49
  Change at Week 24 | -0.8 [-2.54 to 1.00] | 0.9 [-0.94 to 2.72] | 0.1 [-1.66 to 1.91] | 0.3 [-1.53 to 2.05] | -0.1 [-1.50 to 1.35] | -0.8 [-2.14 to 0.60] | -0.5 [-1.82 to 0.88]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.893, Mixed models repeated measures analysis; Adjusted Mean Difference = 0.19, 95% CI 2-sided [-2.62 to 3.00]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.355, Mixed models repeated measures analysis; Adjusted mean difference = 1.33, 95% CI 2-sided [-1.49 to 4.15]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.655, Mixed models repeated measures analysis; Adjusted mean difference = -0.64, 95% CI 2-sided [-3.45 to 2.17]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.719, Mixed models repeated measures analysis; Adjusted mean difference = -0.49, 95% CI 2-sided [-3.20 to 2.21]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.768, Mixed models repeated measures analysis; Adjusted mean difference = 0.41, 95% CI 2-sided [-2.31 to 3.12]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.199, Mixed models repeated measures analysis; Adjusted mean difference = 1.66, 95% CI 2-sided [-0.88 to 4.20]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.483, Mixed models repeated measures analysis; Adjusted mean difference = 0.90, 95% CI 2-sided [-1.62 to 3.41]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.420, Mixed models repeated measures analysis; Adjusted mean difference = 1.03, 95% CI 2-sided [-1.49 to 3.56]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.488, Mixed models repeated measures analysis; Adjusted mean difference = -0.69, 95% CI 2-sided [-2.67 to 1.28]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.694, Mixed models repeated measures analysis; Adjusted mean difference = -0.39, 95% CI 2-sided [-2.36 to 1.58]

11. Secondary Outcome: Percent Change From Baseline in Apolipoprotein AII (ApoAII) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | 8.1 [-14.72 to 30.96] | 18.4 [-4.09 to 40.90] | 8.5 [-13.70 to 30.72] | 8.7 [-14.06 to 31.38] | 5.4 [0.61 to 10.12] | 3.8 [-0.91 to 8.48] | 6.4 [1.82 to 11.08]
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 46 | 43 | 47 | 49
  Percent Change at Week 24 | 5.5 [-15.36 to 26.30] | 15.3 [-5.26 to 35.81] | 2.8 [-17.47 to 23.03] | 8.5 [-12.22 to 29.23] | 0.6 [-2.72 to 3.89] | -1.4 [-4.59 to 1.78] | -0.7 [-3.89 to 2.39]
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.527, Mixed models repeated measures analysis; Adjusted mean difference = 10.29, 95% CI 2-sided [-21.73 to 42.30]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.981, Mixed models repeated measures analysis; Adjusted mean difference = 0.39, 95% CI 2-sided [-31.49 to 32.26]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12; Test type: Superiority or Other; p = 0.974, Mixed models repeated measures analysis; Adjusted mean difference = 0.54, 95% CI 2-sided [-31.72 to 32.80]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.640, Mixed models repeated measures analysis; Adjusted mean difference = -1.58, 95% CI 2-sided [-8.25 to 5.09]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12; Test type: Superiority or Other; p = 0.750, Mixed models repeated measures analysis; Adjusted mean difference = 1.08, 95% CI 2-sided [-5.61 to 7.77]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.509, Mixed models repeated measures analysis; Adjusted mean difference = 9.80, 95% CI 2-sided [-19.41 to 39.01]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.855, Mixed models repeated measures analysis; Adjusted mean difference = -2.69, 95% CI 2-sided [-31.76 to 26.38]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24; Test type: Superiority or Other; p = 0.839, Mixed models repeated measures analysis; Adjusted mean difference = 3.04, 95% CI 2-sided [-26.39 to 32.47]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.392, Mixed models repeated measures analysis; Adjusted mean difference = -1.99, 95% CI 2-sided [-6.57 to 2.59]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24; Test type: Superiority or Other; p = 0.565, Mixed models repeated measures analysis; Adjusted mean difference = -1.33, 95% CI 2-sided [-5.91 to 3.24]

12. Secondary Outcome: Change From Baseline in Total Cholesterol at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 43 | 43 | 46 | 47 | 48 | 50
  Change at Week 12 | -5.6 (29.58) | -35.8 (24.73) | -52.7 (32.67) | -58.6 (32.90) | -0.4 (40.00) | -19.5 (27.39) | -37.6 (43.58)
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Change at Week 24 | -5.5 (28.04) | -31.7 (32.53) | -55.0 (38.67) | -46.9 (33.83) | -6.4 (33.98) | -24.5 (25.86) | -28.6 (33.61)

13. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 43 | 43 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | -2.35 (14.406) | -18.96 (12.299) | -26.45 (14.943) | -31.64 (18.012) | 1.24 (16.624) | -10.51 (15.318) | -19.44 (22.054)
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | -2.31 (13.481) | -16.70 (15.860) | -27.77 (16.993) | -24.31 (16.491) | -1.35 (14.426) | -12.38 (13.365) | -14.61 (17.302)

14. Secondary Outcome: Change From Baseline in Lipoprotein (a) (Lp [a]) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Change at Week 12 | 1.654 (9.8020) | -0.515 (17.6889) | -2.956 (9.9368) | -4.334 (14.3377) | 1.547 (12.0489) | 0.502 (15.1527) | -5.195 (12.9577)
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Change at Week 24 | 1.065 (13.2025) | -1.893 (18.8951) | -3.945 (16.2841) | -3.205 (11.6380) | 2.718 (12.9153) | 2.191 (26.1574) | -3.281 (16.9586)

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) (Lp [a]) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 45 | 44 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | 6.11 (30.573) | 40.43 (333.949) | -11.89 (22.517) | -9.01 (35.644) | 9.28 (33.809) | -0.91 (26.271) | -11.93 (23.893)
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | 8.78 (43.596) | 43.97 (330.964) | -10.18 (26.612) | 0.03 (50.256) | 10.18 (32.604) | -0.79 (25.066) | -5.42 (22.451)

16. Secondary Outcome: Change From Baseline in Very Low Density Lipoprotein (VLDL) Cholesterol at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 42 | 41 | 42 | 45 | 48 | 49
  Change at Week 12 | -12.3 (50.98) | -11.8 (35.82) | -6.0 (46.43) | -20.3 (43.27) | 2.5 (39.66) | -5.8 (38.21) | -12.1 (51.36)
  Change at Week 24: number analyzed (Participants) | 47 | 41 | 42 | 43 | 42 | 46 | 48
  Change at Week 24 | -4.8 (46.55) | -11.5 (49.20) | -12.4 (38.58) | -24.3 (57.43) | -12.1 (40.35) | -15.3 (47.53) | 2.8 (41.81)

17. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein (VLDL) Cholesterol at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 42 | 41 | 42 | 45 | 48 | 49
  Percent Change at Week 12 | 9.62 (71.415) | 2.81 (54.888) | -3.77 (54.845) | -15.61 (36.099) | 17.58 (54.707) | 17.32 (94.238) | 2.16 (80.149)
  Percent Change at Week 24: number analyzed (Participants) | 47 | 41 | 42 | 43 | 42 | 46 | 48
  Percent Change at Week 24 | 20.26 (101.188) | 5.34 (59.092) | -9.78 (39.626) | -13.28 (44.197) | -3.60 (40.646) | 15.72 (142.996) | 33.89 (131.723)

18. Secondary Outcome: Change From Baseline in Triglycerides at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 43 | 44 | 46 | 47 | 48 | 50
  Change at Week 12 | -14.1 (54.92) | -28.7 (76.49) | -17.5 (87.65) | -17.6 (74.45) | 9.0 (66.03) | -9.1 (46.91) | -15.7 (58.22)
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Change at Week 24 | -5.0 (51.01) | -13.0 (100.36) | -25.2 (83.78) | -25.5 (66.92) | -12.0 (45.73) | -20.7 (54.93) | 6.0 (50.52)

19. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 43 | 44 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | -1.17 (42.789) | -5.01 (40.253) | -7.13 (35.229) | -8.93 (50.315) | 13.92 (49.563) | -1.88 (28.283) | -5.91 (39.286)
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | 5.11 (52.717) | 6.49 (51.960) | -10.29 (32.708) | -10.34 (32.992) | -2.01 (29.868) | -7.29 (35.954) | 13.90 (45.386)

20. Secondary Outcome: Change From Baseline in Non-High Density Lipoprotein-Cholesterol (Non-HDL-C) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
milligram per deciliter
  Change at Week 12: number analyzed (Participants) | 47 | 43 | 43 | 46 | 47 | 48 | 50
  Change at Week 12 | -5.7 (26.92) | -37.5 (22.40) | -55.0 (32.75) | -59.6 (33.23) | 0.6 (38.04) | -22.9 (29.05) | -40.7 (44.91)
  Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Change at Week 24 | -5.4 (26.84) | -33.2 (29.21) | -55.9 (38.79) | -47.3 (33.71) | -6.8 (31.49) | -26.3 (22.98) | -28.9 (34.50)

21. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein-Cholesterol (Non-HDL-C) at Week 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percent change
  Percent Change at Week 12: number analyzed (Participants) | 47 | 43 | 43 | 46 | 47 | 48 | 50
  Percent Change at Week 12 | -2.28 (20.234) | -28.34 (15.836) | -38.52 (21.362) | -44.86 (24.258) | 2.76 (20.337) | -17.30 (22.324) | -28.68 (30.857)
  Percent Change at Week 24: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 49
  Percent Change at Week 24 | -2.02 (18.694) | -24.89 (18.938) | -38.02 (23.039) | -34.02 (22.788) | -1.78 (17.145) | -19.39 (17.304) | -19.99 (24.887)

22. Secondary Outcome: Percentage of Participants With Positive Anti-drug (Anti-PF-04950615) Antibodies (ADA)
Description: Participants with titer value greater than or equal to 4.32 nanogram per milliliter were considered positive.
Time Frame: Baseline up to Day 211 for every 28 days groups and Baseline up to Day 225 for every 14 days groups
Population: Analysis set included all participants who received at least 1 dose of PF-04950615.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 51 | 49 | 50 | 51
percentage of participants | 6.0 | 3.9 | 10.2 | 6.0 | 9.8

23. Secondary Outcome: Percentage of Participants With Injection Site Adverse Events
Description: Injection site adverse events included injection site bruising, discomfort, erythema, hemorrhage, induration, inflammation, pain, paresthesia, pruritus, swelling, urticaria, reaction and rash.
Time Frame: Baseline up to Day 211 for 28 days groups and Baseline up to Day 225 for 14 days groups
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 49 | 50 | 51 | 49 | 51 | 50 | 51
percentage of participants | 0 | 4.0 | 0 | 2.0 | 0 | 0 | 2.0

24. Secondary Outcome: Plasma Concentration of PF-04950615 at Week 12 and 24
Time Frame: Week 12, 24
Population: Analysis set included all participants who received at least 1 dose of PF-04950615. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 51 | 49 | 50 | 51
Microgram per milliliter
  Week 12: number analyzed (Participants) | 43 | 41 | 42 | 48 | 49
  Week 12 | 1.0157 (2.09363) | 1.4737 (1.35406) | 2.0516 (2.25916) | 0.5035 (0.53400) | 2.2010 (3.91444)
  Week 24: number analyzed (Participants) | 40 | 42 | 46 | 47 | 49
  Week 24 | 0.7951 (0.78411) | 1.1605 (0.72802) | 1.6500 (2.77210) | 0.3752 (0.41778) | 1.6459 (4.20348)

25. Secondary Outcome: Percentage of Participants With Low Density Lipoprotein-cholesterol Less Than (<) 100, <70, <40 and <25 Milligram Per Deciliter (mg/dL)
Time Frame: Week 12, 24
Population: FAS included all participants who were randomized. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Number analyzed (Participants) | 50 | 50 | 52 | 50 | 51 | 50 | 51
percentage of participants
  Week 12: <100 mg/dL: number analyzed (Participants) | 47 | 44 | 42 | 46 | 46 | 48 | 50
  Week 12: <100 mg/dL | 48.9 | 90.9 | 95.2 | 91.3 | 34.8 | 64.6 | 78.0
  Week 24: <100 mg/dL: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 48
  Week 24: <100 mg/dL | 42.6 | 86.0 | 91.1 | 91.5 | 44.2 | 78.7 | 79.2
  Week 12: <70 mg/dL: number analyzed (Participants) | 47 | 44 | 42 | 46 | 46 | 48 | 50
  Week 12: <70 mg/dL | 4.3 | 50.0 | 66.7 | 78.3 | 0 | 33.3 | 58.0
  Week 24: <70 mg/dL: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 48
  Week 24: <70 mg/dL | 6.4 | 55.8 | 73.3 | 68.1 | 2.3 | 21.3 | 43.8
  Week 12: <40 mg/dL: number analyzed (Participants) | 47 | 44 | 42 | 46 | 46 | 48 | 50
  Week 12: <40 mg/dL | 0.0 | 6.8 | 16.7 | 47.8 | 0 | 8.3 | 32.0
  Week 24: <40 mg/dL: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 48
  Week 24: <40 mg/dL | 0.0 | 4.7 | 22.2 | 17.0 | 0 | 2.1 | 6.3
  Week 12: <25 mg/dL: number analyzed (Participants) | 47 | 44 | 42 | 46 | 46 | 48 | 50
  Week 12: <25 mg/dL | 0.0 | 4.5 | 4.8 | 10.9 | 0.0 | 2.1 | 6.0
  Week 24: <25 mg/dL: number analyzed (Participants) | 47 | 43 | 45 | 47 | 43 | 47 | 48
  Week 24: <25 mg/dL | 0.0 | 0.0 | 4.4 | 2.1 | 0.0 | 0.0 | 2.1
Statistical Analysis 1: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 14.964, 95% CI 2-sided [3.997 to 56.020]
Statistical Analysis 2: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 49.615, 95% CI 2-sided [7.984 to 308.328]
Statistical Analysis 3: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.842, 95% CI 2-sided [3.674 to 44.892]
Statistical Analysis 4: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12, Less than 100 mg/dL; Test type: Superiority or Other; p = 0.010, Regression, Logistic; Odds Ratio (OR) = 3.107, 95% CI 2-sided [1.304 to 7.401]
Statistical Analysis 5: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 12, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.048, 95% CI 2-sided [2.402 to 15.225]
Statistical Analysis 6: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 12.773, 95% CI 2-sided [3.932 to 41.495]
Statistical Analysis 7: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 36.886, 95% CI 2-sided [8.330 to 163.335]
Statistical Analysis 8: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24, Less than 100 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.750, 95% CI 2-sided [5.741 to 75.006]
Statistical Analysis 9: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24, Less than 100 mg/dL; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 6.219, 95% CI 2-sided [2.061 to 18.764]
Statistical Analysis 10: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24, Less than 100 mg/dL; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 6.205, 95% CI 2-sided [2.060 to 18.693]
Statistical Analysis 11: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.703, 95% CI 2-sided [5.752 to 133.423]
Statistical Analysis 12: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 71.177, 95% CI 2-sided [13.783 to 367.564]
Statistical Analysis 13: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 12, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 100.667, 95% CI 2-sided [19.855 to 510.387]
Statistical Analysis 14: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 15: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 24.941, 95% CI 2-sided [6.336 to 98.169]
Statistical Analysis 16: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 80.004, 95% CI 2-sided [18.094 to 353.742]
Statistical Analysis 17: Comparison: Placebo: Every 14 Days vs PF-04950615 150 mg: Every 14 Days; Week 24, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 42.101, 95% CI 2-sided [10.621 to 166.894]
Statistical Analysis 18: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24, Less than 70 mg/dL; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 11.700, 95% CI 2-sided [1.396 to 98.075]
Statistical Analysis 19: Comparison: Placebo: Every 28 Days vs PF-04950615 300 mg: Every 28 Days; Week 24, Less than 70 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 36.841, 95% CI 2-sided [4.527 to 299.817]
Statistical Analysis 20: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12, Less than 40 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 21: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12, Less than 40 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 22: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12, Less than 40 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 23: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24, Less than 40 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 24: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24, Less than 40 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 25: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24, Less than 40 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 26: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 12, Less than 25 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 27: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 12, Less than 25 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 28: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 12, Less than 25 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 29: Comparison: Placebo: Every 14 Days vs PF-04950615 50 mg: Every 14 Days; Week 24, Less than 25 mg/dL; Test type: Superiority or Other; p = 1.000, Regression, Logistic; Odds Ratio (OR) = 1.587
Statistical Analysis 30: Comparison: Placebo: Every 14 Days vs PF-04950615 100 mg: Every 14 Days; Week 24, Less than 25 mg/dL; Test type: Superiority or Other; p < 0.001, Regression, Logistic
Statistical Analysis 31: Comparison: Placebo: Every 28 Days vs PF-04950615 200 mg: Every 28 Days; Week 24, Less than 25 mg/dL; Test type: Superiority or Other; p = 1.000, Regression, Logistic; Odds Ratio (OR) = 0.925

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE. However, what are presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study. Safety analysis set included all participants who received at least 1 dose of study treatment.
Arm/Group | Placebo: Every 14 Days | PF-04950615 50 mg: Every 14 Days | PF-04950615 100 mg: Every 14 Days | PF-04950615 150 mg: Every 14 Days | Placebo: Every 28 Days | PF-04950615 200 mg: Every 28 Days | PF-04950615 300 mg: Every 28 Days
Serious Adverse Events (participants affected / at risk) | 7/49 | 4/50 | 2/51 | 4/49 | 2/51 | 5/50 | 4/51
Other Adverse Events (participants affected / at risk) | 35/49 | 27/50 | 38/51 | 35/49 | 28/51 | 32/50 | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo: Every 14 Days (N=49) | PF-04950615 50 mg: Every 14 Days (N=50) | PF-04950615 100 mg: Every 14 Days (N=51) | PF-04950615 150 mg: Every 14 Days (N=49) | Placebo: Every 28 Days (N=51) | PF-04950615 200 mg: Every 28 Days (N=50) | PF-04950615 300 mg: Every 28 Days (N=51)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exposure via father (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/25 | 0/26 | 0/26 | 0/29 | 0/22 | 0/31 | 0/26 — This event was gender specific.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatic dysplasia (Reproductive system and breast disorders) | 1/25 | 0/24 | 0/26 | 0/21 | 0/29 | 0/19 | 0/25 — This event was gender specific.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: Every 14 Days (N=49) | PF-04950615 50 mg: Every 14 Days (N=50) | PF-04950615 100 mg: Every 14 Days (N=51) | PF-04950615 150 mg: Every 14 Days (N=49) | Placebo: Every 28 Days (N=51) | PF-04950615 200 mg: Every 28 Days (N=50) | PF-04950615 300 mg: Every 28 Days (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 2 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 4 | 5 | 2 | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 5 | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 3 | 1 | 3 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 3 | 2 | 2 | 1
Injection site erythema (General disorders) | 2 | 2 | 4 | 5 | 0 | 4 | 5
Injection site pain (General disorders) | 4 | 4 | 1 | 1 | 2 | 1 | 3
Injection site pruritus (General disorders) | 0 | 0 | 0 | 3 | 0 | 3 | 2
Injection site reaction (General disorders) | 1 | 3 | 1 | 6 | 1 | 1 | 5
Bronchitis (Infections and infestations) | 4 | 2 | 3 | 5 | 3 | 3 | 2
Influenza (Infections and infestations) | 1 | 0 | 2 | 1 | 2 | 1 | 3
Localised infection (Infections and infestations) | 1 | 0 | 3 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 8 | 7 | 5 | 7 | 6 | 6
Sinusitis (Infections and infestations) | 2 | 3 | 3 | 3 | 2 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 5 | 3 | 9 | 5 | 3
Urinary tract infection (Infections and infestations) | 3 | 1 | 5 | 4 | 1 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 1 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3 | 1
Arthalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 6 | 4 | 3 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 2 | 1 | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 3 | 2 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 4 | 1 | 2 | 2 | 1
Headache (Nervous system disorders) | 2 | 2 | 2 | 2 | 1 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 2 | 1 | 1 | 1
Hypertension (Vascular disorders) | 4 | 0 | 2 | 3 | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
There were no limitations or caveats in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results